CLINICAL TRIAL: NCT03809312
Title: The Use of Prophylactic Antibiotics in Endoscopy Sinus Surgery for Chronic Rhinosinusitis With or Without Polyp: A Randomized, Double-blind Clinical Trial
Brief Title: The Use of Prophylactic Antibiotics in Endoscopy Sinus Surgery for Chronic Rhinosinusitis With or Without Polyp
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Simon-Pierre Harvey-Bolduc, ENT resident, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ATBprophylacticCES
Record Dates: First submitted 2019-01-15; First posted 2019-01-18 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Chronic Sinus Infection
Keywords: ESS; Prophylactic antibiotics; Chronic sinus infection
MeSH Terms: interventions — Amoxicillin; Clavulanic Acid

STUDY DESIGN:
Intervention Model Description: During the surgery, 4 groups will be formed as described in the figure below. Patients will be divided according to the presence or absence of polyps at the endoscopy and randomized in one of the 2 groups by the pharmacy of the CHU of Quebec. This will give either a prescription of Clavulin 875 mg per os to be taken twice a day for 10 days, or a placebo of similar visual appearance according to the same dosage
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomisation by the pharmacy, no one in the investigator and the participant will know the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Clavulin group with polyps (Active Comparator): Group who will receive clavulin after the endoscopic sinus surgery in prophylactic and who have polyps in the surgery
  Interventions: Drug: Amoxicillin / Clavulanic acid 875mg / 125mg
- Placebo group with polyps (Placebo Comparator): Group who will receive placebo after the endoscopic sinus surgery in prophylactic and who have polyps in the surgery
  Interventions: Drug: Placebos
- Clavulin group without polyps (Active Comparator): Group who will receive clavulin after the endoscopic sinus surgery in prophylactic and who haven't polyps in the surgery
  Interventions: Drug: Amoxicillin / Clavulanic acid 875mg / 125mg
- Placebo group without polyps (Placebo Comparator): Group who will receive clavulin after the endoscopic sinus surgery in prophylactic and who haven't polyps in the surgery
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Amoxicillin / Clavulanic acid 875mg / 125mg — Amoxicillin / Clavulanic acid 875 mg / 125 mg BID x 10 days
  Arms: Clavulin group with polyps; Clavulin group without polyps
Drug: Placebos — Placebos BID x 10 days
  Arms: Placebo group with polyps; Placebo group without polyps

SUMMARY:
This is a randomized, double-blind clinical trial on the prophylactic use of antibiotics in postoperative endoscopic sinus vs placebo surgery. Patients with chronic rhinosinusitis with or without polyps who have consented to endoscopic sinus surgery according to Canadian practice guidelines may be included in the study after approval by the Research Ethics Board of the University Hospital Center. Quebec and signature of consent.

DETAILED DESCRIPTION:
The severity of the disease will be evaluated preoperatively according to the SNOT-22 score, the visual analogue scale of nasal symptoms, the Lund-Mackay score on the CT-scan and the Modified Lund-Kennedy endoscopic score (sinusoscopy will be recorded). Relevant demographics and medical history of participants will also be collected preoperatively.

The extension of the CES and intraoperative findings will be noted. Patients who have an infection during the procedure (pus with positive culture) will be excluded from the study. During the surgery, 4 groups will be formed as described in the figure below. Patients will be divided according to the presence or absence of polyps at the endoscopy and randomized in one of the 2 groups by the pharmacy of the CHU of Quebec. This will provide either a prescription of Clavulin 875 mg per os twice daily for 10 days, or a placebo of similar visual appearance in the same dosage. A bioabsorbable dressing (NasoPore, Stryker) will be positioned at the mid-meatus level at the end of the procedure. Nasal irrigations of saline solution will be prescribed post-operatively (qid for 1 month) as well as intra-nasal corticosteroids bid after 1 week (usual treatment). The addition of systemic corticosteroids will be left to the judgment of the surgeon, noted and analyzed as a confounding factor.

Follow-up will be done at 2 weeks, 1 month, 3 months and 6 months post-surgery. Patients will have to complete the SNOT-22 quality of life score and the visual similar scale of nasal symptoms at each visit. Sinusoscopy will be recorded at scheduled visits postoperatively. A single blind evaluator (to limit inter-rater differences) will analyze the video recordings to establish the modified Lund-Kennedy endoscopic score for each patient. Middle-meat secretion culture will be performed if pus is present during sinusoscopy and an antibiotic prescribed if needed. The patient will have to fill in a diary of other medications (analgesics, narcotics, anti-inflammatories) as well as a diary of side effects that will be collected at the visit of a post-operative month.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and over able to consent
* Patients with chronic rhinosinusitis and failure to maximal medical treatment
* Endoscopic sinus surgery with at least one of the following: maxillary antrostomy, ethmoidectomy, sphenoidotomy and / or frontal sinusotomy

Exclusion Criteria:

* Antibiotherapy less than 2 weeks before the intervention
* Penicillin allergy
* Inability to establish follow-up
* Open sinus surgery or associated septorhinoplasty (simple septoplasty is not considered an exclusion criterion)
* Immunodeficiency
* Cystic fibrosis of the pancreas
* Pregnancy
* odontogenic sinusitis
* Fungal sinusitis
* Diabetic
* Ciliary dyskinesia
* Sinus neoplasia
* Patient requiring antibiotic prophylaxis for endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2019-08-14 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Modified Lund-Kennedy endoscopic score | 3 months
  The modified Lund-Kennedy score is an endoscopic score that measures sinus involvement during endoscopy. It is divided into 2 nostrils. For each nostril, it has a score of 0 to 2 for the presence of polyp, edema and flow. The score is therefore 0 to 6 for each nostril for a maximum of 12. The higher the score, the more severe is the condition
Quality of life of patients SNOT-22 | 3 months
  The SNOT-22 score is a quality of life score. It contains 22 sinus symptoms. Each of the symptoms is scored from 0 to 5, with 0 being no problem and 5 being a severe problem. The SNOT-22 is a score of 0 to 110, the higher the score, the more severe the disease.

SECONDARY OUTCOMES:
Modified Lund-Kennedy endoscopic score | 1 months
  The modified Lund-Kennedy score is an endoscopic score that measures sinus involvement during endoscopy. It is divided into 2 nostrils. For each nostril, it has a score of 0 to 2 for the presence of polyp, edema and flow. The score is therefore 0 to 6 for each nostril for a maximum of 12. The higher the score, the more severe is the condition
Rate of infection | 3 months
  Evaluate the rate of infection after endoscopic sinus surgery with or without prophylactic antibiotics, defined according to the criteria of acute bacterial rhinosinusitis.
VAS symptoms | 3 months
  The visual analogue scale is a scale containing 6 rhinological symptoms. On a 10 centimeter scale, the patient will write the important of his symptoms, 10 being the maximum and 0 the minimum.
Side effects | 3 months
  Compare side effects when using prophylactic antibiotics after endoscopic sinus surgery for chronic rhinosinusitis versus placebo.
Modified Lund-Kennedy endoscopic score | 6 months
  The modified Lund-Kennedy score is an endoscopic score that measures sinus involvement during endoscopy. It is divided into 2 nostrils. For each nostril, it has a score of 0 to 2 for the presence of polyp, edema and flow. The score is therefore 0 to 6 for each nostril for a maximum of 12. The higher the score, the more severe is the condition
Quality of life of patients SNOT-22 | 1 months
  The SNOT-22 score is a quality of life score. It contains 22 sinus symptoms. Each of the symptoms is scored from 0 to 5, with 0 being no problem and 5 being a severe problem. The SNOT-22 is a score of 0 to 110, the higher the score, the more severe the disease.
Quality of life of patients SNOT-22 | 6 months
  The SNOT-22 score is a quality of life score. It contains 22 sinus symptoms. Each of the symptoms is scored from 0 to 5, with 0 being no problem and 5 being a severe problem. The SNOT-22 is a score of 0 to 110, the higher the score, the more severe the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Simon-Pierre Harvey-Bolduc, Québec, Canada

IPD SHARING:
Plan to Share IPD: No